CLINICAL TRIAL: NCT03489954
Title: Relationship of Deep Cervical Flexor Muscle Endurance With Neck Position Sense and Body Balance in Non-specific Chronic Neck Pain
Brief Title: Relationship of Deep Cervical Flexor Muscle Endurance With Neck Position Sense and Body Balance
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Kübra Karadeniz, Principal Investigator, Dokuz Eylul University
Other Study IDs: 3411-GOA
Record Dates: First submitted 2018-03-25; First posted 2018-04-06 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Neck Pain
Keywords: Chronic Neck Pain; Balance Master; Joint Position Error; Endurance
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-specific chronic neck pain group: In evaluation of participants, endurance of deep cervical flexor muscles will be measured using stabilizer pressure biofeedback unit with cranio-cervical flexion test. Neck position sense of 6-direction (flexion, extension, right-left lateral flexion and right-left rotation) will be measured by CROM device (cervical range of motion device). Body balace will be measured by Balance Master System.
  Interventions: Other: Evaluation
- Healthy group: In evaluation of participants, endurance of deep cervical flexor muscles will be measured using stabilizer pressure biofeedback unit with cranio-cervical flexion test. Neck position sense of 6-direction (flexion, extension, right-left lateral flexion and right-left rotation) will be measured by CROM device (cervical range of motion device). Body balace will be measured by Balance Master System.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — Deep cervical flexor muscle endurance, neck position sense and body balance will be measured.

SUMMARY:
The aims of this research are to investigate relationship of deep cervical flexor muscle endurance with neck position sense and body balance in non-specific chronic neck pain, and to compare the results with healthy individuals.

DETAILED DESCRIPTION:
The investigation will be included 2 groups which include 30 individuals with non-specific chronic neck pain and 30 healthy individuals. In evaluation of participants, endurance of deep cervical flexor muscles will be measured using Stabilizer Pressure Biofeedback Unit with cranio-cervical flexion test. Pressure rise which increases from 20 mmHg to 30 mmHg with 2 mmHg increments will be performed in 5 stages. There are 10 seconds contractions at every stage and these contractions will be made 10 times. Endurance will be calculated by the cumulative performance index with the information obtained from this test. Neck position sense of 6-direction (flexion, extension, right-left lateral flexion and right-left rotation) will be measured by CROM device (cervical range of motion device). Joint position error will be calculated by taking the average of the absolute angular difference by 3 trial for each direction. Body balace will be measured by Balance Master System. Modified clinical test of sensory interaction balance (mCTSIB), limits of stability (LOS), rhythmic weight shift (RWS), unilateral stance (US), walk across (WA) and step/quick turn (SQT) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific chronic neck pain for at least 3 months
* Neck pain is at most 7/10 according to VAS

Exclusion Criteria:

* Musculoskeletal treatment for neck complaints or balance within the last 3 months
* Musculoskeletal disease that may affect balance
* Spine, upper or lower limb fractures or surgical history
* Diagnosis of vestibular disorder
* Diagnosis of neurological or systemic musculoskeletal disease
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals in Dokuz Eylul University Health Campus
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Endurance of deep cervical flexor muscles | Baseline
  Score of cranio-cervical flexion test will be measured by Stabilizer Pressure Biofeedback Unit.

SECONDARY OUTCOMES:
Neck position sense | Baseline
  Joint position error of 6-direction (flexion, extension, right-left lateral flexion and right-left rotation) will be measured by cervical range of motion device (CROM device).
Modified clinical test of sensory interaction balance (mCTSIB) | Baseline
  This test will be measured by Balance Master System.
Limits of stability (LOS) | Baseline
  This test will be measured by Balance Master System.
Rhythmic weight shift (RWS) | Baseline
  This test will be measured by Balance Master System.
Unilateral stance (US) | Baseline
  This test will be measured by Balance Master System.
Walk across (WA) | Baseline
  This test will be measured by Balance Master System.
Step/quick turn (SQT) | Baseline
  This test will be measured by Balance Master System.
Pain | Baseline
  This test will be measured by Visual Analog Scale (VAS) score in activity and rest. VAS has 10-centimeter line corresponding to the amount of pain they experienced. "0" means "no pain" and "10" means "pain as bad as possible".

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi YESILYAPRAK, PhD, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Balçova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No